CLINICAL TRIAL: NCT02491372
Title: A Pilot Study of the Effectiveness of Acceptance and Commitment Therapy With a Post-Upper GI Cancer Population
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit sufficient number of participants in the time available.
Sponsor: Martin Dempster (Other)
Collaborators: Belfast Health and Social Care Trust (Other)
Responsible Party: Sponsor-Investigator, Martin Dempster, Senior Lecturer, Queen's University, Belfast
Organization: Queen's University, Belfast (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B15/01
Record Dates: First submitted 2015-06-05; First posted 2015-07-08 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Acceptance and commitment therapy group
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Comparison (No Intervention): Treatment as usual

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — ACT is a psychological intervention that aims to promote adaptive coping and encourages participants to move their focus away from trying to control emotions to accepting and adapting to them. It is relevant to all patients, not just those who are currently distressed.
  Arms: Intervention

SUMMARY:
This pilot research study aims to assess the effectiveness of an Acceptance and Commitment Therapy (ACT; Hayes Strosahl & Wilson, 2011) group based intervention at improving quality of life (QOL) and increasing Psychological Flexibility with survivors of Upper GI cancer following curative treatment. Participants will be invited to take part in an eight week intervention with outcomes being measured at baseline, midpoint, post-intervention and two month follow up. Outcomes will be compared with a randomised control group who will receive treatment as usual. Research has indicated that this population are under considerable psychological distress however within the UK there are currently no specifically tailored psychological interventions on offer to reduce this distress (Dempster, McCorry, Brennan, Donnelly, Murray & Johnston, 2012).

DETAILED DESCRIPTION:
Design: This pilot study will take the form of a 2 group randomised controlled trial (intervention vs treatment as usual). Measures will be administered at baseline, midpoint, post-intervention and 2 month follow-up.

Setting: Outpatients' clinic. Target population: Adults with oesphagectomy in the previous 3-12 months for oesophageal cancer.

Exclusion Criteria: In receipt of a psychological intervention; have had a reoccurrence of the disease since their surgery; evidence of cognitive impairment impeding ability to engage with the intervention.

Health technology: A group-based acceptance and commitment therapy (ACT) intervention. There will be 2 intervention groups, both of which will receive an 8 week (1.5 hours per week) intervention.

Measurement of costs and outcomes: Participants will be allocated to treatment or control using a randomisation procedure, generated by a statistician outside the research team.

According to the COMET initiative, there are no recommended core outcomes available for use in oesophageal cancer. Work to develop these outcome measures is currently underway and the investigators will contact the authors of this work for the latest updates prior to submitting a full application to ensure that our choice of outcome measures is commensurate with any recommendations they are about to make. In the absence of this work being advanced sufficiently to inform this proposal, the following reliable and valid measures will be used: EORTC Quality of Life Questionnaire and Oesophageal Cancer Module, Acceptance and Action Questionnaire II, which provides a measure of psychological inflexibility, and (secondarily) Depression, Anxiety and Stress Scale.

Sample size: A sample size of 50 (25 per study arm).[42] This will also allow us to estimate a participation rate of 70% to within a 95% confidence interval of ±13%, which will inform the design of the definitive trial.

Current pathway: Patients can seek support for emotional issues from the specialist nurses in the service.

Expertise: Multidisciplinary team including cancer specialist nurses, a service user representative, health economist, statistician, psychologists and with expertise in the intervention to be tested, trials methodology, qualitative and quantitative methods, and research among people with oesophageal cancer

ELIGIBILITY:
Inclusion Criteria:

* Adults diagnosed with Upper GI/ Oesophageal cancer that have undergone an oesphagectomy between three to 12 months previously

Exclusion Criteria:

* Are in receipt of a psychological intervention specifically to deal with the side effects of their oesphagectomy prior to stating the study group.
* Have had a reoccurrence of the disease since their operation
* Show evidence of cognitive impairment which may impede their ability to engage with the intervention.
* Are zero to 3 months post medical intervention to cure their Upper GI/oesophageal cancer (oesphagetomy procedure).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Change in psychological flexibility assessed using the Acceptance and Action Questionnaire II | Pretest, approximately 8 weeks later and then another 3 months later

SECONDARY OUTCOMES:
Change in Depression, anxiety and stress using the Depression Anxiety and Stress Scale 21 | Pretest, approximately 8 weeks later and then another 3 months later
Change in Quality of life using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Oesophageal and Gastric Cancer | Pretest, approximately 8 weeks later and then another 3 months later